CLINICAL TRIAL: NCT05332379
Title: Measurement of Regional Hemodynamic Parameters Before and After Spinal Anesthesia with Doppler USG
Brief Title: Regional Hemodynamic Parameter Changes After Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ruslan Abdullayev, Assist. Prof., Marmara University
Other Study IDs: 09.2021.1406
Record Dates: First submitted 2022-04-11; First posted 2022-04-18 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2023-10

CONDITIONS: Spinal Anesthesia Evaluation
Keywords: Spinal anesthesia; Test; Pulsed Wave Doppler; Sympathectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Diagnostic Test: Pulsed Wave Doppler USG examination — Pulsed Wave Doppler USG examination of the posterior tibial artery on the left or right lower extremity will be performed before spinal anesthesia, at the 5th and 10th minutes after the spinal anesthesia. Blood flow velocities and vessel diameters will be measured.

SUMMARY:
Spinal anesthesia is a regional anesthesia method used for surgical procedures generally involving the lower abdominal area, perineum, and lower extremities. Various tests are performed to evaluate the block level after spinal anesthesia, incluyding pinprick test, cold application, and motor examination. These tests are performed to check whether the pain, sympathetic and motor nerve fibers are affected, respectively, after the block; and good communication with the patient is important here. However, it is extremely difficult to evaluate these tests in pediatric, geriatric, mentally retarded or uncooperative patients.

Sympathectomy can be used as a criterion to evaluate the success of the block that occurs after the spinal anesthesia procedure. Sympathetic nerve fibers are the first to be affected by the block, and the success of the block can be evaluated with the revealed sympathectomy. Sympathectomy in the lower extremities after spinal block increases arterial blood flow. This increase in blood flow can be detected by the Pulsed Wave Doppler feature of USG.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery under spinal anesthesia
* American Society of Anesthesiologists (ASA) I-II physical status

Exclusion Criteria:

* Contraindication for spinal anesthesia
* ASA physical status >II
* Vasoactive drug usage

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients scheduled for elective operation with spinal anesthesia will be recruited for the study. Posterior tibial artery velocities (peak systolic, end-diastolic) and the vessel diameters will be measured via USG Pulsed Wave Doppler mode. Three measurements will be performed: before spinal anesthesia, at the 5th and at the 10th minutes after the subarachnoid injection. The patients' sensory and motor examinations will be performed as well.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2022-04-01 (Actual); Primary Completion 2023-07-20 (Actual); Study Completion 2023-07-20 (Actual)

PRIMARY OUTCOMES:
Arterial velocity changes | At the 5th and 10th minutes after the spinal anesthesia procedure
  Posterior tibial artery velocities (peak systolic, end-diastolic) and vessel diameters will be measured after the spinal anesthesia procedure.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Medicine, Istanbul, Pendik, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided